CLINICAL TRIAL: NCT04849221
Title: Wideband Tympanometry for Monitoring Intracranial Pressure in Adult Patients in Intensive Care, Operated on for an Intracranial Lesion After Traumatic Brain Injury, or With Intracranial Hemorrhage
Acronym: TYMPIC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BOZORG NOURRISSON 2020
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Intracranial Pressure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Head trauma, patient operated on for an intracranial lesion, or other condition (hemorrhagic stroke)
  Interventions: Other: Tympanometry measurement in both ears; Other: Collection of clinical and paraclinical data; Other: Intracranial pressure reading (ICP)
- healthy subjects: No otologic or neurological history
  Interventions: Other: Collection of clinical and paraclinical data; Other: Intracranial pressure reading (ICP)

INTERVENTIONS:
Other: Tympanometry measurement in both ears — Measurement once or twice a day and at every change of more than 10 mmHg in ICP, over the entire period of time that ICP is measured by a probe or DVE
  Groups: Patients
Other: Collection of clinical and paraclinical data — Patient: gender, weight/height, age, etiology of ICP entry, reason for ICP monitoring, presence of external (otoscopy), middle (otoscopy + CT) or internal (CT) ear abnormality, presence of inclusion and non-inclusion criteria, measurement of patient tilt.
  healthy subjects: gender, weight/height, age, presence of abnormality of the external (otoscopy), middle (otoscopy) or internal ear (questioning), presence of inclusion and non-inclusion criteria...
Other: Intracranial pressure reading (ICP) — a single measure

SUMMARY:
Intracranial pressure is usually measured by invasive methods requiring an intracranial sensor. There is no non-invasive monitoring method recognized as a gold standard. Tympanometry would make it feasible to evaluate intracranial pressure through sensitive and specific changes in the energy absorbance of the middle ear. It could represent a non-invasive method of monitoring intracranial pressure.

This is a prospective monocentric longitudinal study. All adult patients in intensive care for head trauma, intracranial hypertension, or after cranial surgery and requiring invasive monitoring of ICP will be included after their non-opposition has been collected.

In a group of 10 controls, multifrequency tympanometry will be performed in the standing position, in the 0° supine position and in the Tredelenburg position at -17°.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Person who did not oppose to their inclusion in the trial
* Head trauma, patient operated on for an intracranial lesion, or other condition (hemorrhagic stroke...) requiring monitoring of ICP by a subdural or epidural sensor.
* Age > 18 years old

Controls:

* Person who did not oppose to their inclusion in the trial
* Age > 18 years old
* No otologic or neurological history.

Exclusion Criteria:

* Person subject to a measure of legal protection (curatorship, guardianship)
* Person under judicial control
* Pregnant, parturient or breastfeeding woman
* Minor
* Fracture of the petrosal bone, abnormality of the bilateral middle or inner ear or canal preventing tympanometry

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head trauma patient operated on for an intracranial lesion or other condition (hemorrhagic stroke)
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2021-08-22 (Actual); Study Completion 2021-08-22 (Actual)

PRIMARY OUTCOMES:
Volume of the ear canal as a function of intracranial pressure | Approximately on the 10th day
Width between conductance peaks of tympanometry at 2kHz as a function of intracranial pressure | Approximately on the 10th day
Middle ear resonance frequency as a function of intracranial pressure | Approximately on the 10th day

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourogne, Dijon, France